CLINICAL TRIAL: NCT04637490
Title: Patellar Resurfacing in Total Knee Arthroplasty Leads to Better Isokinetic Performance and Higher Clinical Scores
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Deniz CANKAYA, Associate Professor, Gulhane Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-17-1414
Record Dates: First submitted 2020-11-09; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Knee Osteoarthritis
Keywords: patellar resurfacing; isokinetic testing
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patellar resurfacing (Experimental): patellar resurfacing in TKA
  Interventions: Device: patellar component
- non-resurfacing (No Intervention): non-resurfacing TKA

INTERVENTIONS:
Device: patellar component — patellar resurfacing
  Arms: patellar resurfacing

SUMMARY:
For decades there have been concerns about patellar resurfacing (PR) in total knee arthroplasty (TKA) and the individual preference of the surgeon is still the main determinant of whether or not resurfacing is applied. According to preference, surgeons can be categorized in 3 main groups of those who usually, selectively or rarely resurface. The aim of this prospective, randomized, controlled study to is compare the isokinetic performance and clinical outcome of TKAs with PR and without PR.

DETAILED DESCRIPTION:
Patients undergoing TKA for primary osteoarthritis of the knee are randomly assigned to either the PR or non-PR groups. The differences between groups with respect to age, BMI, gender, and preoperative Knee Society Score (KSS), and isokinetic performance are evaluated. Patients are evaluated at postoperative 3, 6, and 12 months with KSS and at 6 months and 1 year with isokinetic measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 55 to 80 years
* unilateral primary osteoarthritis

Exclusion Criteria:

* bilateral osteoarthritis
* inflammatory arthritis
* post-traumatic osteoarthritis
* previous knee surgery
* neuromuscular diseases

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
isokinetic test | Change from preoperative isokinetic test results at 6th months and 12th months isokinetic test results
  isokinetic test during extension and flexion of the knee

SECONDARY OUTCOMES:
Knee Society Score (KSS): It has two different subscales: Knee and Function 100-80: Excellent 79-70:Good 69-60:Fair below 60:Poor | Change from preoperative KSS results at 3rd months, 6th months and 12th months KSS results
  Knee Society Score (KSS)

CONTACTS AND LOCATIONS:
Overall Officials: Deniz CANKAYA, Assoc.Professor, Principal Investigator — Gulhane Teaching and Research Hospital
Locations (1):
- Gulhane Teaching and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No